CLINICAL TRIAL: NCT02155244
Title: Common Bile Duct Stone Management: What Have we Learned?
Acronym: CBDS
Status: Completed | Type: Observational
Sponsor: Ospedale Regionale di Mendrisio (Other)
Responsible Party: Principal Investigator, Luca Regusci, MD, Ospedale Regionale di Mendrisio
Other Study IDs: LR-1234
Record Dates: First submitted 2014-05-19; First posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Common Bile Duct Stones
Keywords: CBDS; ERCP; Dindo-Clavien classification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Common bile duct stones: Common bile duct stones traeted with ERCP
- CBDS: treated with ERCP combined with surgery

SUMMARY:
In unfit elderly people with comorbid disease leaving the gallbladder in situ is justified after ERCP treatment. Cholangitis is more present in elderly people. The purpose of this study is to determine leaving the gallbladder in situ does not reduce the morbidity rate after ERCP for common bile duct stones(CBDS), especially in patients with cholangitis.

DETAILED DESCRIPTION:
The prevalence of gallstone disease increases with age, and as many as one third of women and one fifth of men over the age of 60 years have gallstones. The quoted prevalence of CBDS in patients with symptomatic gallstones varies, but probably lies between 10 and 20%. In Europe and Northern America 8 to 20% of cases of cholelithiasis is complicated by presence of common bile duct stones (CBDS) during cholecystectomy. When ductal stones do become symptomatic the consequences are often serious and can include pain, partial or complete biliary obstruction, cholangitis, hepatic abscesses or pancreatitis. Recent guidelines for the treatment of CBDS recommend that in patients with symptoms and clinical evaluation suggesting ductal stones as a cause, stones should be extracted if possible, except in selected patients that have contraindications (e.g high risks patients, refusal of endoscopic or operative treatment).

Many different approaches are currently being used for the management of bile duct calculi. These strategies differ considerably in terms of technical complexity, sensitivity, specificity, effectiveness, and cost. Where initial assessment suggests a high probability of CBDS, then it is reasonable to proceed directly to ERCP if this is considered the treatment of choice. Intraoperative cholangiography with selective intraoperative or postoperative ERCP is a strategy than routine preoperative ERCP, unless the presence of common bile duct stones (CBD) is almost certain. Current data does not suggest clear superiority of any one approach with regard success, mortality, morbidity and cost-effectiveness. In unfit elderly people with comorbid disease leaving the gallbladder in situ is justified after ERCP treatment. Cholangitis is more present in elderly people. Leaving the gallbladder in situ does not reduce the morbidity rate after ERCP for CBDS, especially in patients with cholangitis

All 101 patients with symptomatic and suspected CBD stones admitted to Surgical Department of "Ospedale Regionale di Mendrisio" from january 2006 to december 2013 were evaluated retrospectively for study eligibility. Patients were followed for the duration of hospital stay, the median hospital stay was 9 days.

From our Hospital informatic system, information on age, sex, length of hospital stay, and procedures undertaken during hospital admissions for patients with biliary diagnoses were retrieved. Initial patient evaluations consisted of history and physical examinations and serum analyses for inflammatory parameters, bilirubin, alkaline phosphatase, transaminase, and amylase. Previous history of jaundice or acute pancreatitis was recorded. In addition, right upper quadrant abdominal sonograms and CT scan were obtained for the determination of cholelithiasis and CBD diameter. The diagnosis of cholangitis was based on presence of clinical evidence of infection in patients with biliary obstruction in the form of jaundice or hyperbilirubinemia.

In our institution, patients with cholelithiasis, a CBD stones at US examination, and liver enzyme elevation, without clinical evidence of cholecystitis or biliary pancreatitis underwent ERCP, endoscopic sphincterotomy, and endoscopic clearance of CBD stones before laparoscopic cholecystectomy (LC). In patients with acute cholangitis, a dilated common bile duct on US, the first treatment was also ERCP. Patients with cholelithiasis, CBD and intrahepatic bile duct (IHBD) dilatation, and liver enzyme elevation, in the presence of cholecystitis, biliary pancreatitis, or apparent resolving symptomatic choledocholithiasis underwent further evaluation with magnetic resonance imaging(MR), and these patients underwent therapeutic ERCP when choledocholithiasis was demonstrated by MR, whereas patients whose MR did not detect choledocholithiasis underwent LC with intraoperative cholangiography (IOC). When we found CBD during LC, an ERCP was performed in the same operating time ("rendez-vous") or post operatively.

Endoscopic retrograde cholangiopancreatography(ERCP) with papillotomy was performed in patients with confirmed common bile duct stones(CBDS) by a single gastroenterologist.

In our Hospital, the procedure is performed in radiological room that contains x-ray equipment. We use a Olympus® duodenalendoscope TJF-145 for ERCP, Erbe® system for papillotomy diathermy, and Lithotriptor® if stone crushing is necessary. The patient is in prone position under general anesthesia. When performing endoscopic stone extraction the endoscopist has the support of a technician or radiologist who can assist in fluoroscopic screening and an additional endoscopy assistant/nurse to manage guide wires.

The relationship between ERCP and surgery was assessed by dividing the patients into 2 groups: patients who had ERCP without cholecystectomy (Group 1), patients who had ERCP + cholecystectomy (Group 2). Endpoint was to detect difference in age, indication (cholangitis and lithiasis), morbidity, effectiveness and success of CBD clearance in different groups.

ELIGIBILITY:
Inclusion Criteria:

- Patients with common bile duct stones (CBDS)

Exclusion Criteria:

Ages: 18 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2006-01; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Post-operative complications according to Clavien-Dindo classification | During patients hospitalization (median hospital stay was 9 days)